CLINICAL TRIAL: NCT03999931
Title: The Second Affiliated Hospital, Zhejiang University
Brief Title: Study on the Difference of Plasma microRNA Expression in Patients With Genetic Susceptibility to Mental Disorders
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-058
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2016-06

CONDITIONS: Plasma microRNA in Patients With Genetic Susceptibility to Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- schizophrenia with positive symptoms: schizophrenia with positive symptoms
- schizophrenia with negative symptoms: schizophrenia with negative symptoms
- bipolar disorder: bipolar disorder
- depression: depression
- panic disorder: panic disorder
- obsessive-compulsive disorder: obsessive-compulsive disorder
- control

SUMMARY:
Schizophrenia (Schizophrenia,Sc), biphasic affective disorder (Bipolar disorder,BPD), major depression (major depressive disorder,MDD), anxiety disorder (Anxiety disorder,An) and other mental disorders have obvious family aggregation, with heritability of 60 -90%. This kind of common mental illness seriously affects the psychosomatic health and quality of life of patients, and places a great mental and economic burden on the society and family. At present, the diagnosis of mental illness is mainly based on clinical symptoms. With the development of molecular biology, genomics has become a new way to study mental illness. MicroRNA (miRNA) is a class of eukaryotic endogenously non-coding single-stranded RNA, which can regulate gene expression by binding to specific mRNA or regulating the protein translation process of specific mRNA. MiRNA widely exists in plasma and serum, and the type and quantity of miRNA in plasma and serum change with different physiological and disease conditions. It is reported that the expression profile of miRNA in brain tissue of schizophrenia is significantly different from that of normal subjects. In addition, the study found that the specific miRNA detected in peripheral blood can directly reflect the condition of the disease, which may use miRNA in peripheral blood as a clinical biological marker. In order to detect the expression of various miRNA in plasma, high throughput miRNA chip detection has become the first choice for primary screening. In this study, the investigators intend to detect the difference of miRNA expression in peripheral blood of different types of schizophrenia by high throughput miRNA chip, and analyze the correlation between them. It is hoped to provide the basis for the diagnosis and occurrence and development of clinical psychotic patients.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria of DSM- V (see attached page for details); there is no history of blood transfusion within 1 month.

Exclusion Criteria:

Physical and nervous system diseases such as brain trauma; history of mental illness such as mental retardation; history of alcohol abuse and drug abuse.

Ages: 21 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From 2014 to 2016, 28 patients with mental disorders were enrolled in the second affiliated Hospital of Zhejiang University, aged 21 -66 years, with an average age of 42.0 years.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The expression of mir-4687-3p in patients with PD is different from that in normal subjects. | July, 2016
  The expression of mir-4687-3p in patients with PD is different from that in normal subjects.

IPD SHARING:
Plan to Share IPD: Undecided